CLINICAL TRIAL: NCT05119712
Title: Terbinafine Treatment of Axial Spondyloarthropathy
Acronym: FUN
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study stopped due to poor recruitment.
Sponsor: Oregon Health and Science University (Other)
Collaborators: The Malassezia Foundation (Unknown)
Responsible Party: Principal Investigator, Atul Deodhar, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00021565
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Ankylosing Spondylitis; Axial Spondyloarthritis; Psoriatic Spondylitis; Spondylitis Secondary to Inflammatory Bowel Disease; Axial Spondyloarthopathy
Keywords: fungus, malassezia, microbiome
MeSH Terms: conditions — Spondylitis, Ankylosing; Axial Spondyloarthritis | interventions — Terbinafine; Clinical Laboratory Techniques; Urinalysis

STUDY DESIGN:
Intervention Model Description: Subjects will receive either terbinafine 500 mg or placebo for 16 weeks and then crossed over to the opposite therapy for another 16 weeks.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo to Drug (Active Comparator): Subjects will begin treatment on placebo then crossover to study drug.
  Interventions: Drug: Terbinafine Tablets; Diagnostic Test: Laboratory Testing
- Drug to Placebo (Active Comparator): Subjects will begin treatment on study drug then crossover to placebo.
  Interventions: Drug: Terbinafine Tablets; Diagnostic Test: Laboratory Testing

INTERVENTIONS:
Drug: Terbinafine Tablets — 500mg oral terbinafine or placebo daily
  Other Names: Lamisil
Diagnostic Test: Laboratory Testing — Laboratory testing at screening, baseline, week 8, 16, 24 and 32.
  Other Names: Blood work
Diagnostic Test: Laboratory Testing — Subjects with the potential to become pregnant will have a baseline urine pregnancy test prior to starting study drug.
  Other Names: Urinalysis

SUMMARY:
This is a pilot study to determine if further research is warranted to assess if anti-fungal therapy is an effective adjunctive treatment for axial spondyloarthropathy

DETAILED DESCRIPTION:
The purpose of this trial is to determine if terbinafine is an effective therapy for ankylosing spondylitis. Benefit will be determined by a reduction of the BASDAI by two or more.

The primary endpoint is the BASDAI at the completion of 16 weeks of terbinafine versus the BASDAI at the start of the trial and at the completion of the placebo. The secondary endpoint with the percent of patients whose BASDAI improves by two or more while on terbinafine (week 16) versus the percent of subjects with a similar improvement after 16 weeks of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 and older of either sex will be included.
* Subjects must be willing and able to provide informed consent.
* Subjects must have been diagnosed with ankylosing spondylitis, axial spondyloarthritis, psoriatic spondylitis or spondylitis secondary to inflammatory bowel disease by a physician and must be willing to request records to validate the diagnosis.
* Subjects must complete a symptom questionnaire called a BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) and must have a score of four or above to indicate active disease and the potential to improve.
* Subjects must agree to remain on a stable treatment regimen for their joint disease for the duration of the trial and for one month before the study begins.
* Subjects must be willing to provide stool samples and be willing to have routine lab studies every 8 weeks during the duration of the study.

Exclusion Criteria:

* Pregnant or lactating women will not be included.
* Subjects must not be allergic or intolerant to terbinafine.
* Subjects must not be taking medications that have the potential for serious interactions with terbinafine. These drugs include desipramine, cimetidine, fluconazole, cyclosporine and rifampin.
* Subjects must not have taken antibiotics within 3 months of starting the study drug and collecting the baseline stool specimen.
* Subjects with the following blood dyscrasias will not be included:

Hemoglobin <9g/dL or Hematocrit <30% White blood cell count <3.0 K/cu mm Absolute neutrophil count <1.2 K/cu mm Platelet count <100 K/cu mm Subjects with an estimated GFR ≤50 ml/min Subjects with a total bilirubin, AST, or ALT more than 1.5 times the upper limit of normal at screening.

* Severe, progressive, or uncontrolled chronic liver disease including fibrosis, cirrhosis, or recent or active hepatitis.
* History of any lymphoproliferative disorder such as Epstein Barr virus (EBV) related lymphoproliferative disorder, history of lymphoma, leukemia, or signs and symptoms suggest of current lymphatic disease.
* Current malignancy or history of malignancy, with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ.
* Have or have had an opportunistic infection (e.g., herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis and aspergilloma, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening.
* Have a known infection with human immunodeficiency virus (HIV)
* Have current signs and symptoms of systemic lupus erythematosus, or severe, progressive, or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac (New York Heart Association class III or IV), neurologic, or cerebral diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in BASDAI score | 16 weeks
  BASDAI score after the completion of 16 weeks of terbinafine treatment versus the BASDAI score after 16 weeks on placebo. Benefit is defined by a reduction of BASDAI score of 2 or more.

CONTACTS AND LOCATIONS:
Overall Officials: Atul Deodhar, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.

REFERENCES:
- [Background] Reveille JD, Witter JP, Weisman MH. Prevalence of axial spondylarthritis in the United States: estimates from a cross-sectional survey. Arthritis Care Res (Hoboken). 2012 Jun;64(6):905-10. doi: 10.1002/acr.21621. Epub 2012 Jan 24. PMID 22275150
- [Background] Goie The HS, Steven MM, van der Linden SM, Cats A. Evaluation of diagnostic criteria for ankylosing spondylitis: a comparison of the Rome, New York and modified New York criteria in patients with a positive clinical history screening test for ankylosing spondylitis. Br J Rheumatol. 1985 Aug;24(3):242-9. doi: 10.1093/rheumatology/24.3.242. PMID 3160423
- [Background] Asquith M, Rosenbaum JT. The interaction between host genetics and the microbiome in the pathogenesis of spondyloarthropathies. Curr Opin Rheumatol. 2016 Jul;28(4):405-12. doi: 10.1097/BOR.0000000000000299. PMID 27152700
- [Background] Laurence M, Asquith M, Rosenbaum JT. Spondyloarthritis, Acute Anterior Uveitis, and Fungi: Updating the Catterall-King Hypothesis. Front Med (Lausanne). 2018 Apr 5;5:80. doi: 10.3389/fmed.2018.00080. eCollection 2018. PMID 29675414
- [Background] Mielants H, Veys EM, De Vos M, Cuvelier C, Goemaere S, De Clercq L, Schatteman L, Elewaut D. The evolution of spondyloarthropathies in relation to gut histology. I. Clinical aspects. J Rheumatol. 1995 Dec;22(12):2266-72. PMID 8835560
- [Background] Maillet J, Ottaviani S, Tubach F, Roy C, Nicaise-Rolland P, Palazzo E, Dieude P. Anti-Saccharomyces cerevisiae antibodies (ASCA) in spondyloarthritis: Prevalence and associated phenotype. Joint Bone Spine. 2016 Dec;83(6):665-668. doi: 10.1016/j.jbspin.2015.10.011. Epub 2016 Mar 15. PMID 26992953
- [Background] Gross O, Gewies A, Finger K, Schafer M, Sparwasser T, Peschel C, Forster I, Ruland J. Card9 controls a non-TLR signalling pathway for innate anti-fungal immunity. Nature. 2006 Aug 10;442(7103):651-6. doi: 10.1038/nature04926. Epub 2006 Jul 12. PMID 16862125
- [Background] Zhernakova A, Festen EM, Franke L, Trynka G, van Diemen CC, Monsuur AJ, Bevova M, Nijmeijer RM, van 't Slot R, Heijmans R, Boezen HM, van Heel DA, van Bodegraven AA, Stokkers PC, Wijmenga C, Crusius JB, Weersma RK. Genetic analysis of innate immunity in Crohn's disease and ulcerative colitis identifies two susceptibility loci harboring CARD9 and IL18RAP. Am J Hum Genet. 2008 May;82(5):1202-10. doi: 10.1016/j.ajhg.2008.03.016. Epub 2008 Apr 24. PMID 18439550
- [Background] Pointon JJ, Harvey D, Karaderi T, Appleton LH, Farrar C, Stone MA, Sturrock RD, Brown MA, Wordsworth BP. Elucidating the chromosome 9 association with AS; CARD9 is a candidate gene. Genes Immun. 2010 Sep;11(6):490-6. doi: 10.1038/gene.2010.17. Epub 2010 May 13. PMID 20463747
- [Background] Ruutu M, Thomas G, Steck R, Degli-Esposti MA, Zinkernagel MS, Alexander K, Velasco J, Strutton G, Tran A, Benham H, Rehaume L, Wilson RJ, Kikly K, Davies J, Pettit AR, Brown MA, McGuckin MA, Thomas R. beta-glucan triggers spondylarthritis and Crohn's disease-like ileitis in SKG mice. Arthritis Rheum. 2012 Jul;64(7):2211-22. doi: 10.1002/art.34423. PMID 22328069
- [Background] Takahata Y, Sugita T, Hiruma M, Muto M. Quantitative analysis of Malassezia in the scale of patients with psoriasis using a real-time polymerase chain reaction assay. Br J Dermatol. 2007 Oct;157(4):670-3. doi: 10.1111/j.1365-2133.2007.08090.x. Epub 2007 Jul 19. PMID 17634085
- [Background] Limon JJ, Tang J, Li D, Wolf AJ, Michelsen KS, Funari V, Gargus M, Nguyen C, Sharma P, Maymi VI, Iliev ID, Skalski JH, Brown J, Landers C, Borneman J, Braun J, Targan SR, McGovern DPB, Underhill DM. Malassezia Is Associated with Crohn's Disease and Exacerbates Colitis in Mouse Models. Cell Host Microbe. 2019 Mar 13;25(3):377-388.e6. doi: 10.1016/j.chom.2019.01.007. Epub 2019 Mar 5. PMID 30850233
- [Background] Babu PR, Pravin AJS, Deshmukh G, Dhoot D, Samant A, Kotak B. Efficacy and Safety of Terbinafine 500 mg Once Daily in Patients with Dermatophytosis. Indian J Dermatol. 2017 Jul-Aug;62(4):395-399. doi: 10.4103/ijd.IJD_191_17. PMID 28794551
- [Background] Chapman SW, Pappas P, Kauffmann C, Smith EB, Dietze R, Tiraboschi-Foss N, Restrepo A, Bustamante AB, Opper C, Emady-Azar S, Bakshi R. Comparative evaluation of the efficacy and safety of two doses of terbinafine (500 and 1000 mg day(-1)) in the treatment of cutaneous or lymphocutaneous sporotrichosis. Mycoses. 2004 Feb;47(1-2):62-8. doi: 10.1046/j.1439-0507.2003.00953.x. PMID 14998402